CLINICAL TRIAL: NCT03090360
Title: Growth of Infants Fed a New Term Infant Formula With a Prebiotic
Brief Title: Growth of Infants Fed a New Term Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 16.07.INF
Record Dates: First submitted 2017-03-08; First posted 2017-03-24 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Healthy
Keywords: Healthy babies; Infant formula; Growth
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo comparator (Control) (Placebo Comparator): Starter infant formula with a probiotic and without a prebiotic. Volumes of feed depend on age, weight and appetite.
  Interventions: Dietary Supplement: Infant formula (CF)
- Experimental Formula (Test) (Experimental): Starter infant formula with a probiotic and prebiotic. Volumes of feed depend on age, weight and appetite.
  Interventions: Dietary Supplement: Infant Formula (EF)
- Breastfed reference group (No Intervention): Breastfed reference group

INTERVENTIONS:
Dietary Supplement: Infant formula (CF) — Formula-fed infants will be randomly assigned to receive one of the study formulas (CF or EF) orally, ad libitum, each day from Study Day 1 until Study Day 180, for a treatment duration of approximately 180 days.
  Arms: Placebo comparator (Control)
Dietary Supplement: Infant Formula (EF) — Formula-fed infants will be randomly assigned to receive one of the study formulas (CF or EF) orally, ad libitum, each day from Study Day 1 until Study Day 180, for a treatment duration of approximately 180 days.
  Arms: Experimental Formula (Test)

SUMMARY:
To evaluate the growth of healthy term infants fed an experimental infant formula with a prebiotic, a commercial control infant formula with a probiotic, but without a prebiotic and human breast milk

DETAILED DESCRIPTION:
Multisite, double-blind, randomized, controlled clinical trial. The purpose of the study is to determine if infants fed a standard infant formula with a prebiotic have a weight gain in line with infants fed a standard starter infant formula without a prebiotic.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed and dated
2. Infants whose parent(s)/Legally Authorized Representative (LAR) have reached the legal age of majority in Belgium
3. Infants whose parent(s)/LAR are willing and able to comply with scheduled visits, and the requirements of the study protocol.
4. Infants whose parent(s)/LAR are able to be contacted directly by telephone throughout the study.
5. Infants whose parent(s)/LAR have a working freezer.
6. Healthy term, singleton infant at birth.
7. At enrollment visit, post-natal age ≤ 14 days (date of birth = day 0).
8. At enrollment, birth weight ≥ 2500g and ≤ 4500g.
9. For formula-fed group, infant of parent(s)/LAR who have previously made the decision to formula feed their infant at the time of enrollment.

Exclusion Criteria:

1. Infants with conditions requiring infant feedings other than those specified in the protocol.
2. Infants receiving complementary foods or liquids.
3. Infants who have a medical condition or history that could increase the risk associated with study participation or interfere with the interpretation of study results.
4. Infants who are presently receiving or have received prior to enrollment medications that could interfere with the interpretation of study results.
5. Infants or infants whose parent(s)/LAR who in the Investigator's assessment cannot be expected to comply with the protocol or with study procedures.

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 349 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
Growth | 120 days
  Growth (weight gain velocity)

SECONDARY OUTCOMES:
Growth | Every month up to 6 months of age
  Other growth outcomes will be compared to the World Health Organization 2006 Growth Standards and by treatment group
Stool patterns (3-day GI symptom and behavior diary - stool frequency and stool consistency) | Every month up to 6 months of age
  Stool patterns (3-day GI symptom and behavior diary - stool frequency and stool consistency)
GI tolerance (3-day GI symptom and behavior diary - including GI symptoms, GI-related behaviors, and milk intake) | Every month up to 6 months of age
  GI tolerance (3-day GI symptom and behavior diary - including GI symptoms (frequency and amount of spitting-up/vomiting, and frequency of flatulence), GI-related behaviors (duration of crying and fussiness, sleeping, and the frequency of excessive crying episodes), and milk intake)
Fecal microbiota composition and diversity (16S rRNA sequencing and qPCR) | Every month up to 4 months of age
  Fecal microbiota composition, diversity, and abundance
Fecal markers (pH, fecal organic acids, and protein markers of gut health) | Every month up to 4 months of age
  Fecal markers (pH, fecal organic acids, and protein markers of gut health)
Gene expression (infant exfoliated and microbial cell gene expression by shotgun sequencing) | Up to 3 months of age
  Gene expression (infant exfoliated and microbial cell gene expression by shotgun sequencing)
Adverse events / Morbidity | 180 days
  Adverse events / Morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Alliet, Principal Investigator — Kinderartsen Huis 5
Locations (7):
- Belgium (5):
  - Algemeen Stedelijk Ziekenhuis Aalst, Aalst
  - UZ Brussel, Brussels
  - Kinderartsen Huis5, Hasselt
  - Clinique Ste Elisabeth, Namur
  - CHwapi, Tournai
- Italy (2):
  - Fondazione Istituto di Ricovero e Cura a Carattere Scientifico Ca' Granda, Ospedale Maggiore Policlinico, Milan
  - AOUP "Paolo Giaccone", Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alliet P, Vandenplas Y, Roggero P, Jespers SNJ, Peeters S, Stalens JP, Kortman GAM, Amico M, Berger B, Sprenger N, Cercamondi CI, Corsello G. Safety and efficacy of a probiotic-containing infant formula supplemented with 2'-fucosyllactose: a double-blind randomized controlled trial. Nutr J. 2022 Feb 22;21(1):11. doi: 10.1186/s12937-022-00764-2. PMID 35193609